CLINICAL TRIAL: NCT00936988
Title: A Multicenter, Open-label Extension Study to Assess the Long-term Safety and Efficacy of an Oral Calcimimetic Agent AMG 073 (Cinacalcet) in Primary Hyperparathyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20000159
Record Dates: First submitted 2009-06-04; First posted 2009-07-10 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Hyperparathyroidism, Primary
Keywords: Hyperparathyroidism, Primary; cinacalcet
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Cinacalcet

ARMS (1):
- cinacalcet (Experimental)
  Interventions: Drug: cinacalcet

INTERVENTIONS:
Drug: cinacalcet — Subjects began open-label treatment with 30 mg cinacalcet twice daily (BID) at the start of the current study. The study consisted of 2 phases planned to total approximately 4¾ years: a 12-week dosetitration phase (visits at weeks 2, 3, 4, 6, 9, and 12) during which 1 possible dose increase of cinacalcet from 30 mg BID to 50 mg BID could occur at week 6, and a maintenance phase (week 12 to 234; visits approximately every 4 weeks until week 24 and approximately every 14 weeks thereafter) during which doses also could be titrated. After July 2004, because of a change in dose strengths, the daily doses used in the study were 30 and 60 mg BID with the option to reduce to 30 mg once daily (QD), if necessary. Ongoing subjects receiving 50 mg BID were switched at that time to 60 mg BID.

SUMMARY:
This multicenter, open-label, single-arm, extension study was designed to evaluate long-term tolerability, safety, and efficacy of cinacalcet. Subjects were enrolled immediately after they completed the parent study, 990120. All subjects began treatment with 30 mg cinacalcet twice daily (BID), with dose adjustments made per protocol-specified guidelines. The study consisted of 2 consecutive phases that occurred in the following order: a dose-titration phase lasting 12 weeks and a maintenance phase lasting approximately 4½ years.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed the parent study 990120
* Agreed to use highly effective (in the opinion of the principal investigator) contraceptive measures throughout the study
* Were able to comprehend and were willing to give written informed consent for participation in the study

Exclusion Criteria:

* Pregnant or breast-feeding
* Had a psychiatric disorder that interfered with the understanding and giving of informed consent or compliance with protocol requirements
* Had any other condition that reduced the chance of obtaining data (eg, known poor compliance)
* Participating in another investigational study at the time of study entry
* Had any unstable medical condition, defined as having been hospitalized within 28 days before day 1, or otherwise unstable in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2000-11; Primary Completion 2005-06 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Nature, frequency, severity, and relationship to treatment of adverse events | 234 weeks

SECONDARY OUTCOMES:
Calcium levels and plasma iPTH during the maintenance phase | 234 weeks
Percentage changes in BMD from baseline of the parent study to each measurement time point and absolute BMD values, as assessed by DXA scans of proximal femur, lumbar spine (L1-L4), forearm, and total body scans | 234 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Peacock M, Bolognese MA, Borofsky M, Scumpia S, Sterling LR, Cheng S, Shoback D. Cinacalcet treatment of primary hyperparathyroidism: biochemical and bone densitometric outcomes in a five-year study. J Clin Endocrinol Metab. 2009 Dec;94(12):4860-7. doi: 10.1210/jc.2009-1472. Epub 2009 Oct 16. PMID 19837909
- [Derived] Peacock M, Bilezikian JP, Bolognese MA, Borofsky M, Scumpia S, Sterling LR, Cheng S, Shoback D. Cinacalcet HCl reduces hypercalcemia in primary hyperparathyroidism across a wide spectrum of disease severity. J Clin Endocrinol Metab. 2011 Jan;96(1):E9-18. doi: 10.1210/jc.2010-1221. Epub 2010 Oct 13. PMID 20943783
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com